CLINICAL TRIAL: NCT06174402
Title: Fenofibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cholangitis
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Ying (Other)
Responsible Party: Sponsor-Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY-20232219-C-1
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fenofibrate-ursodesoxycholic acid（UDCA） (Experimental): Fenofibrate 200 mg/day and UDCA 13-15mg/kg/day for 12 months
  Interventions: Drug: Fenofibrate; Drug: UDCA
- Placebo-UDCA (Placebo Comparator): 1 tablet/ day and UDCA 13-15mg/kg/day for 12 months
  Interventions: Drug: Placebo; Drug: UDCA

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 200 mg/day
  Arms: Fenofibrate-ursodesoxycholic acid（UDCA）
Drug: Placebo — 1 tablet/ day
  Arms: Placebo-UDCA
Drug: UDCA — UDCA 13-15mg/kg/day

SUMMARY:
The main objectives of the study were to assess the effects of fenofibrate on serum alkaline phosphatase, as a composite endpoint and on safety in participants with primary biliary cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

* Must have provided written informed consent
* Age 18-75 years;
* BMI 17-28 kg/m2
* Male or female with a diagnosis of PBC, by at least two of the following criteria:

  1. History of alkaline phosphatase（ALP） above upper limit of normal（ULN） for at least six months;
  2. Positive Anti-mitochondrial antibody (AMA) titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies;
  3. Documented liver biopsy result consistent with PBC.
* Incomplete response to UDCA defined by 1 x ULN< ALP <= 1.67 x ULN
* Taking UDCA for at least 6 months (stable dose for ≥ 3 months) prior to Day 0

Exclusion Criteria:

* History or presence of other concomitant liver diseases.
* ALT or AST > 5×ULN, total bilirubin（TBIL） > 3×ULN.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Allergic to fenofibrate or ursodeoxycholic acid.
* Taking hepatotoxic drugs (e.g., dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than 2 weeks within 6 months, and long-term hormonal users.

Recurrent variceal bleeding, poorly controlled hepatic encephalopathy or refractory ascites.

* Patients with a history of severe cardiac, cerebrovascular, renal, respiratory disease or functional failure, and psychiatric disorders (including those due to alcohol and drug abuse).
* Creatinine >1.5×ULN and creatinine clearance <60 ml/min.
* Currently using statins (such as pravastatin, fluvastatin, and simvastatin), other fibrates (such as gemfibrozil and bezafibrate), and drugs structurally similar to fenofibrate (like ketoprofen).
* Planned to receive an organ transplant or an organ transplant recipient.
* Needing Liver transplantation within 1 year according to the Mayo Rick score.
* Any other condition(s) that would compromise the safety of the subject or compromise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with biochemical response | 48 weeks
  The normalisation of Alkaline Phosphatase

SECONDARY OUTCOMES:
Percentage of patients having biochemical response | 4, 12, 24 and 36weeks
  The normalisation of Alkaline Phosphatase at 4, 12, 24, and 36 weeks
Assessment of the pruritus | 4, 12, 24, 36, and 48 weeks
  Change From Baseline in Pruritus as Assessed by Visual Analogue Scale (VAS) Total Score for Fatigue and Pruritus. (0-10, higher scores mean a worse outcome)
Assessment of the fatigue | 4, 12, 24, 36, and 48 weeks
  Change From Baseline in Fatigue as Assessed by Visual Analogue Scale (VAS) Total Score for Fatigue and Pruritus. (0-10, higher scores mean a worse outcome)
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of creatinine, blood urea nitrogen, alanine aminotransferase and aspartate aminotransferase
Survival without transplantation and hepatic impairment | 48 weeks
  Occurrence of ascites, variceal bleeding, hepatic encephalopathy, liver-transplantation, or death

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The second hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing Second Hospital, Nanjing, Jiangsu
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Xijing Hospital, Xi'an, Shaanxi
  - Yan'an University Affiliated Hospital, Yan’an, Shanxxi
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Peking Union Medical College Hospital, Beijing